CLINICAL TRIAL: NCT04809233
Title: Expanded Access to Tipifarnib
Status: Available | Type: Expanded Access
Sponsor: Kura Oncology, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Expanded Access to Tipifarnib
Record Dates: First submitted 2021-03-18; First posted 2021-03-22 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: HRAS Mutations or Peripheral T Cell Lymphoma (PTCL)
Keywords: Lymphoma; T-Cell; Peripheral; Non-Hodgkin; HRAS; Peripheral T-cell
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral; Lymphoma | interventions — tipifarnib

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Tipifarnib

SUMMARY:
Requests for single patient expanded access to tipifarnib may be considered for adult patients with HRAS mutations or peripheral T Cell Lymphoma (PTCL).

To request access, use Responsible Party contact information provided in this record.

Expanded access for tipifarnib is only available in the United States.

ELIGIBILITY:
Inclusion/Exclusion Criteria:

Diagnosed with HRAS-mutant carcinomas or peripheral T Cell Lymphoma (PTCL).

Adult, ages 18+.

Have exhausted appropriate standard treatments without success and no comparable or satisfactory alternative treatment is available or exists to treat the disease or condition.

Is ineligible for participation in any ongoing clinical study of the investigational drug, which includes lack of access due to geographic limitations.

Meets any other pertinent medical criteria for access to the investigational drug, as established by the Kura Oncology

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult